CLINICAL TRIAL: NCT05819060
Title: The Efficacy and Safety of The Fuzuloparib Combination With Bevacizumab in Maintenance Treatment for Platinum-Sensitive Recurrent Ovarian Cancer
Brief Title: The Efficacy and Safety of The Fuzuloparib Combination With Bevacizumab
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhong Zheng MD, Professor, Director of Gynecologic Oncology, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-02-3121
Record Dates: First submitted 2023-03-19; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Recurrent Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fuzuloparib Combination with Bevacizumab (Experimental): Fuzuloparib 150mg/bid ; Bevacizumab 7.5mg/kg，d1，Q3W
  Interventions: Drug: Fuzuloparib Combination with Bevacizumab

INTERVENTIONS:
Drug: Fuzuloparib Combination with Bevacizumab — For the first 6 patients, if DLT≤33.3%, Fuzuloparib 150mg/bid will be used for follow-up research; if DLT>33.3%, Fuzuloparib will be used for follow-up research at 100mg/bid; Bevacizumab 7.5mg/kg, d1, Q3W.

SUMMARY:
The study will be a Prospective, Single-arm, Phase Ⅱ Clinical Study. This study intends to explore the efficacy and safety of Fuzuloparib combined with bevacizumab in the maintenance treatment of patients with platinum-sensitive ovarian cancer. The progression-free survival, OS, and safety were evaluated based on RECIST V1.1.

DETAILED DESCRIPTION:
Due to the lack of effective predictive molecular markers in the maintenance treatment phase, it is difficult to assess the effectiveness of maintenance treatment. This project plans to collect blood and urine from subjects before maintenance treatment, during relapse, and for follow-up molecular marker exploration research.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with platinum-sensitive recurrent ovarian cancer confirmed by pathology or histology;
2. Patients who have previously received platinum-based chemotherapy and had a recurrence interval of > 6 months before the last platinum-based chemotherapy;
3. Patients who have previously received bevacizumab and did not experience progression within 3 months during the use of bevacizumab;
4. Patients who have previously received PARP inhibitors and did not experience progression within 12 months during the use of PARP inhibitors;
5. The patient achieved a complete or partial response after the last platinum-based chemotherapy;
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
7. The patient has a life expectancy of at least 3 months and sufficient organ function;
8. The patient has sufficient bone marrow reserves and organ function, including a creatinine clearance rate of 45 mL/min calculated using the standard Cockcroft and Gault formula;
9. The patient voluntarily agrees to participate in this study and signs an informed consent form.

Exclusion Criteria:

1. Patients who are known to be allergic or intolerant to chemotherapy drugs or their excipients and cannot swallow medication;
2. Patients who have undergone major surgery within 28 days prior to enrollment;
3. Patients with central nervous system metastases or a history of seizures within the past 12 months;
4. Uncontrolled hypertension: systolic blood pressure ≥180mmHg, diastolic blood pressure ≥90mmHg;
5. NYHA functional class ≥ III;
6. Patients with severe, uncontrolled systemic diseases;
7. Patients who have received any other investigational drug treatment or participated in any other clinical trials within 30 days prior to enrollment in this study;
8. Pregnant or lactating patients, or patients who cannot guarantee effective contraception during the study treatment period;
9. Patients with poorly controlled neurological or psychiatric disorders or mental illness, poor compliance, and inability to cooperate or describe treatment response;
10. Patients judged by the investigator to be unsuitable for participation in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-04-30 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | approximately 1.5 years
  according to RECIST v1.1

SECONDARY OUTCOMES:
Overall survival (OS) | Up to approximately 1.5 years
  according to RECIST v1.1
Adverse Events (AEs) | From the first drug administration to within 30 days for the last treatment dose]
  According to CTCAE V5.0 criteria, During the trial, the adverse event record form should be truthfully filled in, including the occurrence time, severity, correlation with study treatment, duration, measures taken and outcome of the adverse event.

OTHER OUTCOMES:
Exploration of molecular markers | Up to approximately 1.5 years
  Through the analysis of serum and urine proteomics and metabolomics, predictive PFS markers were screened,for example,CA 125, ctDNA

CONTACTS AND LOCATIONS:
Overall Officials: Zhong Zheng, Ph.D, Principal Investigator — Department of Gynecologic Oncology, Fudan University Shanghai Cancer
Locations (1):
- Fudan University Shanghai Cancer Cente, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Data is available per require after approved by ethics broad